CLINICAL TRIAL: NCT02757274
Title: Prospective Registry for Patients Undergoing Surgery for Male Stress Urinary Incontinence in Multiple European Centres
Brief Title: Prospective Registry for Patients Undergoing Surgery for Male Stress Urinary Incontinence
Acronym: SATURN
Status: Active, not recruiting | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: EAU-RF 2016-01
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urologic Surgical Procedure; Male
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a prospective collection of pre-defined parameters on the treatment of male stress urinary incontinence by an artificial urinary sphincter (AUS) and male sling. The data collection will be undertaken from multiple centers in Europe. The participation will be by open invitation to all members of the Female & Functional Section of the EAU (ESFFU) along with other urologists undertaking these procedures. There will be a call via the European Association of urology (EAU) to all European Urologists to register for database entry. There will be no restriction on the number of patients enrolled as long as they are consecutive. The aim is to have a long term collection of the data set from as many centers as possible. An initial assessment for the robustness of the data collection will be undertaken at 3 months by a nominated steering committee. However, the first clinical evaluation of the data collected will commence at 1 year by the steering committee. Thereafter, the evaluations will be performed after every 2 years.

DETAILED DESCRIPTION:
STATISTICS

1. Number of Participants:

   Investigators anticipate to recruit 1000 patients from at least 25-30 European Centers and prospectively collect data from 100 - 200 patients per year. Statistical analysis will be performed on the total number of participants. Based on the available literature, we anticipate an average cure rate of 50% for AUS and for male slings an average cure rate of 65% at the end of study.

   With an estimated sample size of 700 patients treated with Artificial Urethral Sphincter (AUS) and 300 patients with a male sling, and taking into account an attrition rate of 10-15%, we will be able to detect a 50% cure rate with 6% on either side of the 95% Confidence Interval for AUS (proportion 0,50 with 95% Confidence Intervals: 0,44-0,56) and a 65% cure rate for patients treated with male slings (proportion 0,65 with 95% Confidence Intervals: 0,57-0,74).
2. Statistical Analysis:

No adjustment procedures or imputations of missing data will take place.

2.1 Patient characteristics: Patient characteristics as age, weight, length, etc. will be summarized using descriptive statistics - the number of patients with non-missing data, mean, standard deviation, median, minimum and maximum will be presented for continuous outcomes, and the number and percentage of patients in each category will be presented for categorical outcomes. A subgroup analysis by Device subtype will be carried out.

2.2 Primary endpoint analyses: Cure rate will be the main endpoint of the study, and is defined as urinary continence with no need for use of pads or the use of 1 light security pad. The cure rate after 10 years of study follow up will be calculated together with its 95% Confidence Intervals, for the total patient group as well as for each device subtype.

2.3 Secondary endpoints analyses: Time being Incontinence-free will be a secondary endpoint of the study, and is defined as the interval from the date of regaining continence after surgery to the date of incontinence. Continence is defined as no pad use or one light security pad per 24 hours use. Patients who die will be censored at time of death. Overall time being incontinence-free will be presented using the Kaplan-Meier curve, for the total patient group as well as for each device subtype.

Time being revision-free will be another endpoint of the study, and is defined as the interval from the date of surgery to the date of revision. Patients who die will be censored at time of death. Overall time being revision-free will be presented using the Kaplan-Meier curve, for the total patient group as well as for each device subtype.

The results of questionnaires ICIQ Male LUTS Questionnaire SF and EQ-5D-5L will be analysed comparing baseline with 12 weeks post-surgery and the yearly follow up results for the whole group and for the device subgroups. Further, complications (and SADE's), pain and symptoms during and post-surgery and other post-operative data will be evaluated in the device subgroups.

2.4 Prognostic factors: Univariable and multivariable analysis will be carried out to identify clinical and surgical variables that correlate with (in)continence or revisions for each of the device subtypes.

STUDY CONDUCT CONSIDERATIONS

A research co-coordinator will be available in each center for obtaining Ethics Committees (ECs) approval and to deliver logistics of patient screening, follow-up visits, data collection and data entry into the electronic Case Report Form (eCRF).

1. Regulatory and Ethical Considerations:

   Prior to initiation of a study site, the research co-coordinator will obtain approval from the appropriate regulatory agency and ECs to conduct the study in accordance with applicable country-specific regulatory requirements. The study will be conducted in accordance with applicable subject privacy requirements.
2. Recruitment and Consent:

A patient information sheet and consent form will be available and translated in the local language. This form will state that data will be processed anonymously and handled according to local data protection laws. In case a patient is eligible, the physician will verbally inform the patient about this registry and its purpose. The patient will also receive a written patient information sheet in the local language explaining the registry. The patient will be given ample opportunity to ask any questions he might have. The patient will be given as much time as needed to consider his participation in this registry. If a patient agrees to participate, the informed consent form will be signed prior to registration of the patient data.

ADMINISTRATIVE ASPECTS AND PUBLICATION

1. Handling and Storage of Data and Documents:

   All items as described in the protocol will be entered into an eCRF. The physician will guarantee that all team members or other persons involved in the center will respect the confidentiality of any information concerning the registry patients. All parties involved in this registry will maintain strict confidentiality to assure that neither the person nor the family privacy of a patient participating in the registry is violated. Likewise, the appropriate measures shall be taken to avoid the access of non-authorized persons to the registry data. Data will be made anonymous and extracts of the anonymized data will be accessible for reporting and statistical analyses. The processing of the personal data on the patients taking part in this registry, and in particular regarding data concerning consent, shall comply with the local law on the privacy and with the European Directive on the Privacy of data (95/46/EC).
2. Site Audit:

   Site audits will be conducted by the European Association of Urology Foundation for Urological Research (EAU RF) or another designated third party in approximately 5-10% of the sites. To avoid fraud, spot check monitoring and source data verification will be conducted to identify if a patient really exists and if the data entered in the database is retrieved from real patient files and has been transferred correctly.
3. Project Database:

   For the purpose of the study, the data will be stored in a central database held by ESFFU under the umbrella of EAU RF. The investigator or a qualified employee will enter all relevant patient data into a web based electronic Data Capture system. Data checks, programmed in the data capture system, use predefined rules for range or consistency with other data fields in the registry. Data will also be checked for accuracy and correctness by data-managers of the EAU RF according to internal procedures. The site will be capable of modifying the data to assure accuracy with source documentation. At the end of the study, EAU RF will archive the study data in accordance with internal procedures. Specific instructions for use of the eCRF system will be included in the training material provided to the investigational site.
4. Amendments:

   Amendments are changes made to the registry protocol. Amendments will be notified or submitted for approval to the Ethical Committee (EC) as required according to local law.
5. Annual Progress Report:

   According to local requirements, the sponsor will submit a summary of the progress of the registry to the participating physicians and research coordinators for submission to the local ECs (if required) in each country once a year. Information will be provided on the date of inclusion of the first patient, numbers of patients included and numbers of patients that have completed the registry, issues, and amendments.
6. End of Registry Report:

   According to local requirements, the sponsor or physician will notify the Competent Authority (CA), the Central Ethical Committee (CEC) and local ECs of the end of the study. The registry will end after such decision is taken by ESFFU and EAU RF. In case the registry is ended, the sponsor or physician will notify the CA/CEC and local ECs (if required), including the reasons for the premature termination. Within one year after the end of the registry, the sponsor will submit a final registry report with the results of the registry, including any publications/abstracts of the registry, to the CA/CEC and local EC (if required).
7. Steering Committee:

A Steering Committee was assembled, consisting of urologist key opinion leaders in the field of reconstructive surgery and physicians/scientists with clinical and methodological expertise. The Steering Committee is responsible for the assignment of National Coordinators. Each participating country has one National Coordinator who has been selected by the Steering Committee. The Steering Committee will convene once or twice a year.

ELIGIBILITY:
Inclusion Criteria:

* Male patient undergoing surgery for stress incontinence by AUS or male sling.
* Participant is willing and able to complete the questionnaires and give informed consent for participation in the study.

Exclusion Criteria:

* Participating center is unable to contribute consecutive patients.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients undergoing surgery for treatment of stress urinary incontinence by AUS or male sling
Sampling Method: Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 10 years after surgery
  Cure rate will be the main endpoint of the study, and is defined as urinary continence with no need for use of pads or the use of 1 light security pad. The cure rate after 10 years of study follow up will be calculated together with its 95% Confidence Intervals, for the total patient group as well as for each device subtype.

OTHER OUTCOMES:
Time being incontinence-free | 10 years post surgery
  Incontinence-free rate will be a secondary endpoint of the study, and is defined as the interval from the date of surgery to the date of incontinence recurrence. Patients who die will be censored at time of death. Overall time of being incontinence free will be presented using the Kaplan-Meier curve, for the total patient group as well as for each device subtype.
Time being revision-free | 10 years post surgery
  Time being revision-free will be another endpoint of the study, and is defined as the interval from the date of surgery to the date of revision. Patients who die will be censored at time of death. Overall time being revision-free will be presented using the Kaplan-Meier curve, for the total patient group as well as for each device subtype.
Complications | At year 1, year 3, year 5, year 7, year 10
  Number of patients with complications such as: urinary retention (yes or no (Y/N)), scrotal hematoma (Y/N), perineal pain (Y/N), hematuria (Y/N), or other local or general problems (Y/N) will be presented in a tabular format.
Change in quality of life versus baseline (pre-surgery) | At week 12, year 1, and then yearly up to and including year 10.
  The change in quality of life compared with baseline (pre-surgery) will be reported at week 12, year 1, and then yearly up to and including year 10.
Change in the results of the incontinence questionnaire versus baseline (pre-surgery) | At week 12, year 1, and then yearly up to and including year 10.
  The change in the results of the incontinence questionnaire compared with baseline (pre-surgery) will be reported at week 12, year 1, and then yearly up to and including year 10.
Number of patients with postoperative specific events related to the surgical procedure or the sling / prosthesis (e.g. pump/reservoir/cuff failure (Y/N), erosion of the device through the skin (Y/N) or urethra (Y/N)). | At year 1, year 3, year 5, year 7, year 10
  Number of patients with these specific types of events will be presented in a tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Rizwan Hamid, MD, Principal Investigator — Dept of NeuroUrology, London Spinal Injuries Unit, HA7 4LP London, Middlesex, UK; John Heesakkers, MD, Principal Investigator — Dept. of Urology, MUMC, Maastricht, the Netherlands; Frank Van der Aa, MD, Principal Investigator — Dept. of Urology, University Hospital Leuven, Belgium; Nikesh Thiruchelvam, MD, Principal Investigator — Dept. of Urology, CUH-Addenbrooke's Hospital; Wim Witjes, MD, PhD, Study Director — EAU Research Foundation
Locations (28):
- Belgium (5):
  - University Hospital Antwerpen, Antwerp
  - University Hospital Gent, Ghent
  - Jessa Ziekenhuis campus Salvator, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Thomayer Hospital, Prague, Czechia
- Helsinki University Hospital, Helsinki, Finland
- Germany (3):
  - University Medical Center Hamburg Eppendorf, Hamburg
  - Universitätsmedizin Mainz, Mainz
  - University Münster, Münster
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
- Netherlands (2):
  - UMC Radboud, Nijmegen
  - University Medical Center Utrecht, Utrecht
- Norway (2):
  - Universitetssykehuset Nord-Norge, Narvik
  - Oslo University Hospital, Rikshospitalet, Oslo
- Spain (10):
  - Germans Trias i Pujol Universitary Hospital, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - University Hospital La Fe, Valencia
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Guy's Hospital, London
  - Royal National Orthopaedic Hospital, Stanmore

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may share anonymized individual data with residents/urologist interested to analyze and publish the results of the registry

REFERENCES:
- [Result] Heesakkers J, Martens F, Thiruchelvam N, Witjes W, Caris C, Kats J, Hamid R, Van der Aa F; EAU Research Foundation SATURN Study Group. Results at 1 Year from SATURN, A European, Prospective, Multicenter Registry for Male Stress Urinary Incontinence Surgery. Eur Urol Focus. 2024 Sep;10(5):818-825. doi: 10.1016/j.euf.2024.04.003. Epub 2024 Apr 15. PMID 38627124
- [Result] Martens F, Heesakkers J, Van der Aa F, Thiruchelvam N, Witjes W, Caris C, Kats J, Hamid R; EAU Research Foundation SATURN Registry Study Group. SATURN: A European, Prospective, Multicentre Registry for Male Stress Urinary Incontinence Surgery. Eur Urol Open Sci. 2023 Oct 6;57:91-97. doi: 10.1016/j.euros.2023.09.011. eCollection 2023 Nov. PMID 38020526
- [Result] Thiruchelvam N, Heesakkers J, Hamid R, Martens F, der Aa FV, Witjes W, Caris C, Kats J; European Association of Urology Research Foundation SATURN Registry Study Group. SATURN: A Multinational, Multicentre, Prospective Surgical Registry for Male Urinary Incontinence Surgery Across Europe with Planned 10-year Follow-up. Eur Urol Focus. 2025 Mar;11(2):187-189. doi: 10.1016/j.euf.2025.03.004. Epub 2025 Mar 20. PMID 40118692
- See also: EAU Research Foundation website — https://uroweb.org/eau-research-foundation-eau-rf